CLINICAL TRIAL: NCT05679843
Title: Characteristics and Prognosis of STEMI Patients Undergoing Primary PCI According to Coronary Occlusion Physiopathogeny and/or Atherosclerotic Burden
Brief Title: Clinical Characteristics and Prognosis of STEMI Patients Undergoing Primary Percutaneous Coronary Angioplasty and Angiographic Data
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Batric POPOVIC, MD,PhD, Central Hospital, Nancy, France
Other Study IDs: CentralHNF number 2022PI183
Record Dates: First submitted 2022-12-24; First posted 2023-01-11 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
Keywords: STEMI, Gensini,
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gensini score (GS) provides valuable information on severity and prognosis of coronary artery disease (CAD). We aim to evaluate the relationship between the severity of CAD determined by the GS and short and long term of ST-elevation myocardial infarction (STEMI) patients undergoing primary percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with STEMI underwent primary PCI within 24 hours after first symptoms

Exclusion Criteria:

Patients with STEMI 24 hours after first symptoms Pregnant patient <18 years old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with STEMI underwent primary PCI within 24 hours after first symptoms in our hospital
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-06-07 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Composite outcome including all cause death and re myocardial infarction | 6 years

SECONDARY OUTCOMES:
ST resolution on ECG after primary PCI | 1 hour

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Popovic B, Varlot J, Humbertjean L, Sellal JM, Pace N, Hammache N, Fay R, Eggenspieler F, Metzdorf PA, Camenzind E. Coronary Embolism Among Patients With ST-Segment-Elevation Myocardial Infarction and Atrial Fibrillation: An Underrecognized But Deadly Association. J Am Heart Assoc. 2024 May 21;13(10):e032199. doi: 10.1161/JAHA.123.032199. Epub 2024 May 14. PMID 38742522